CLINICAL TRIAL: NCT04869748
Title: A Randomized Controlled Trial Study of Perfetti Method on Upper Extremity Spasticity of Stroke Patient
Brief Title: Perfetti Method on Upper Extremity Spasticity of Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MURA2018/441
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Stroke Syndrome Sequela Spasticity
Keywords: Upper extremity spasticity; stroke; Perfetti method; passive stretching exercise
MeSH Terms: conditions — Stroke | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: single blind randomized controlled trial study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): After recruitment, signed inform consent and allocation, researcher collected demographic data of each participant. First outcome assessment was done before session. Participants received a 15-minute session of Perfetti method on affected elbow flexor.Immediate after session, last outcome assessment was collected.
  Interventions: Other: Perfetti method
- control group (Active Comparator): After recruitment, signed inform consent and allocation, researcher collected demographic data of each participant. First outcome assessment was done before session. Participants received a 15-minute session of Passive stretching on affected elbow flexor.Immediate after session, last outcome assessment was collected.
  Interventions: Other: passive stretching

INTERVENTIONS:
Other: Perfetti method — * Participant was blindfolded, while lying flat in a quiet and comfortable room.
  * Participants received a 15-minute session of Perfetti method on affected elbow flexor.
  * Participants were asked to concentrate on the position of their elbows.
  * Protocol has 4 steps of training starting from 2 positions; full flexion and full extension 3 positions; full flexion, elbow flexion 90 degree and full extension 4 positions; full flexion, elbow flexion 110-140 degree, elbow flexion 45-60 degree and full extension 5 positions; full flexion, elbow flexion 110-140 degree, elbow flexion 90 degree, elbow flexion 45-60 degree and full extension of elbow.
  * After therapist passively moved elbow joint to a position, participant guessed the position of his/her elbow. If the answers were correct consecutively for 10 times, the therapist increased the number of positions according to the protocol.
  Other Names: cognitive sensorimotor training therapy
  Arms: experimental group
Other: passive stretching — * Participant was blindfolded, while lying flat in a quiet and comfortable room.
  * Each participant received gentle passive stretching of elbow flexor and maintained in full elbow extension position for 15 minutes.
  Arms: control group

SUMMARY:
This study objective is to study the immediate effect of Perfetti Method in reducing spasticity of upper extremity in stroke patients at the Department of Physical Medicine,Faculty of Medicine Ramathibodhi Hospital, Thailand. Participants were randomized into experimental group who received therapy according to the Perfetti method, and controlled group who underwent passive stretching exercise. Duration of treatment was 15 minutes for every case, regardless of the treatment. Evaluation of spasticity immediately before and after treatment according to Modified Tardieu scale (MTS) and Modified Ashworth Scale (MAS) by same blinded assessor.

DETAILED DESCRIPTION:
* This study was a single center, single-blind randomized controlled trial study conducted in Thailand during June 2018 and September 2019.
* After approval by Human Research Ethics Committee, Faculty of Medicine Ramathibodi Hospital, Mahidol University, stroke patients with spasticity of upper extremity at the Department of Rehabilitation Medicine, Faculty of Medicine Ramathibodhi Hospital were recruited.
* Participants were assigned to experimental group and control group by researcher using computer randomization.
* Outcome assessor was blinded to the allocations.
* Demographic data including gender, ages, type of stroke, hemiparesis side, time since stroke, duration of upper limb spasticity, Brunnstrom stage of upper extremity, joint proprioception of elbow joint, Barthel index, spasticity impact score, and current treatment (conventional physical therapy, antispastic medication, botulinum toxin/ Phenol injection) were collected. A simplified questionnaire was used to determine spasticity impact score.
* All therapy sessions were conducted by the same PMR residence, who was trained by an experienced occupational therapist for 1 session and further practiced under supervision for 10 sessions.
* The primary outcome was the improvement of the angle of muscle reaction (R1 angle) in Modified Tardieu Scale (MTS).
* The secondary outcomes were the number of participants with improvement of quality of muscle action in MTS ≥1 and the number of participants with improvement of Modified Ashworth Scale (MAS) ≥1.
* Sample size was calculated using delta change of R1 angle of MTS in 10 subjects pilot study, with alpha = 0.05 and beta = 0.1. The total number of sample size is 7 subjects per group, 14 subjects in total.
* In Experimental group, each participant received a 15-minute session of Perfetti method on affected elbow flexor. Participant was blindfolded, while lying flat in a quiet and comfortable room. Participants were asked to concentrate on the position of their elbows. Protocol has 4 steps of training as shown in Table 1, starting from 2 positions of elbow and ending with 5 positions. After therapist passively moved elbow joint to a position, participant guessed the position of his/her elbow. If the answers were correct consecutively for 10 times, the therapist increased the number of positions according to the protocol.
* In control group, each participant received gentle passive stretching of elbow flexor and maintained in full elbow extension position for 15 minutes.
* For statistical analysis, program SPSS version 21 was used to calculate mean and standard deviation (mean±SD) for continuous variables, and percent and median for categorical variables. Paired T-test and independent T-test were used to compared result in the same group and between groups, respectively. Results were considered significant when p <0.05. The difference in quality of muscle reaction of MTS and MAS was deemed meaningful if the reduction was ≥ 1 level.

ELIGIBILITY:
Inclusion Criteria:

1. stroke confirmed by history, physical examination and imaging
2. having spastic elbow flexors MAS ≥ 2
3. full range of motion (ROM) of elbow from 0-150 degree
4. Montreal cognitive assessment (MOCA) score ≥ 23
5. having had problem from spasticity
6. age ≥ 18 years old
7. given written informed consent to participate

Exclusion Criteria:

1. having been treated with Perfetti method
2. previous soft tissue release of involved elbow flexor
3. having wound or inflammation on treatment area
4. unstable medical condition
5. other conditions affecting tone of elbow flexor, e.g. nerve injury
6. not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
angle of muscle reaction (R1 angle) in Modified Tardieu Scale (MTS) | immediate after intervention
  R1 angle in MTS post-session(degree) minus R1 angle in MTS pre-session. Outcome was report in degree, from 0 to 180 degree. Higher value is better outcome.

SECONDARY OUTCOMES:
quality of muscle action in MTS | immediate after intervention
  Number of participants with improvement of quality of muscle action in MTS ≥1. Higher number is better outcome.
  Quality of muscle reaction in MTS is an ordinal scale to assess spasticity, consist of 6 levels, 0, 1, 2, 3, 4 and 5. The worst level of spasticity is 5 and the best level is 0. The improvement of quality of muscle reaction means change in level of quality of muscle reaction from higher to lower ≥1 level .
Modified Ashworth Scale (MAS) | immediate after intervention
  Number of participants with improvement of Modified Ashworth Scale (MAS) ≥1 level. Higher number of participants is better outcome.
  MAS is an ordinal scale to assess spasticity, consist of 6 levels, 0, 1, 1+, 2, 3 and 4. The worst level of spasticity is 4 and the best level is 0. The improvement of MAS means change in level of MAS from higher to lower ≥1 level .

CONTACTS AND LOCATIONS:
Overall Officials: Pimchanok Tuakta, MD, PMR, Principal Investigator — Department of rehabilitation medicine, Faculty of Medicine Ramathibodi Hospital
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand